CLINICAL TRIAL: NCT02326623
Title: Distraction to Reduce Pain and Distress: A Randomized Controlled Trial of Children Undergoing Intravenous Placement in the Pediatric Emergency Department
Brief Title: Distraction to Reduce Pain and Distress in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050791
Record Dates: First submitted 2014-10-10; First posted 2014-12-29 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2017-02

CONDITIONS: Children Requiring IV Placement
MeSH Terms: interventions — Osteogenesis, Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iPad distraction (Experimental): The intervention will be the use of an iPad that will include a selection of child-appropriate games. We will select popular, age-appropriate items to include on the iPad, chosen based on the most current online consumer ratings. Children and parents will be able to select their choice of distraction and can change their selection as desired during the course of the procedure. These choices will be recorded for study purposes.
  Interventions: Other: distraction
- standard care (Other): The control group will receive standard care, which generally includes the use of topical anesthetic cream.
  Interventions: Other: topical anesthetic cream

INTERVENTIONS:
Other: distraction — distraction using an iPad with a selection of child-appropriate games
  Arms: iPad distraction
Other: topical anesthetic cream — standard care is to use a topical anesthetic cream at the site of planning IV access
  Arms: standard care

SUMMARY:
Many medical procedures aimed at helping children can cause them pain and distress. If children have certain levels of pain or distress, it can have long lasting negative effects. The emergency department can be a very stressful place for children and their parents. There are also many procedures that children may have in the emergency department that can cause pain and distress. These include procedures such as needle pokes, stitches, or setting a broken bone. Two common methods of managing a child's pain in the emergency department are drugs and distraction. Drugs are not always practical and may come with unwanted side effects. Distraction is often used by parents or health professionals to help children deal with pain and stress. Distraction can lower the child's pain and distress by moving their attention from the painful experience, for example a needle poke, to a more positive feeling such as watching a movie, playing a game, or listening to music. This study will test if iPads are useful to help lower pain and distress for children (ages 6 to 11 years) who are visiting an emergency department and need an intravenous line put in. The results from this study could be important for many children receiving medical care, as distraction is safe and the use of iPads is enjoyable for many children.

DETAILED DESCRIPTION:
Setting and Study Period: The study will be conducted in the ED of the Stollery Children's Hospital. Patient recruitment is projected to begin in October 2014 and continue to March 2015.

Study Design and Population: The study will be a RCT; the primary outcomes will be the child's self-reported pain and observed behavioural distress. The population is children, ages 6 to 11 years, attending a pediatric ED and requiring IV placement.

Recruitment: Research assistants (RAs) will identify patients attending the ED between the ages of 6 and 11 years. A RA will be on-site from approximately 14:00 to 22:00 daily to identify children who require IV placement; this time corresponds with peak visits requiring IV placements based on data collected in the ED at the Stollery Children's Hospital in team members' previous studies. For those who require IV placement, the RA will further assess child eligibility based on the inclusion / exclusion criteria outlined below. If the child is eligible, the RA will explain the study and invite the parent and child to participate. After obtaining written, informed consent from the parent and assent from the child, the RA will open a prepared randomization envelope and assign the child to one of the two intervention arms. The RA will ask one parent or caregiver for each child to participate and complete all relevant questionnaires.

Baseline Assessment: After informed consent/assent is obtained, the RA will gather information from the parent on baseline demographic variables (e.g., gender, age), presenting signs and symptoms (e.g., chief complaint), and previous history with ED visits and IV placement.

Randomization, Allocation, and Blinding of Study Treatment: Randomization method: A statistician will prepare the randomization sequence using appropriate software and prepare the envelopes. Allocation will be concealed from the RAs, ED staff, child and parent until consent/assent has been obtained. The statistician will maintain the randomization code which will not be broken until data analysis is complete. Allocation: After receiving informed consent/assent, the RA will open the next envelope in a series of consecutively labeled, sealed, opaque envelopes. These will be kept in a secured location in the ED research office. Blinding: Due to the nature of the intervention, it will not be possible to blind the children, parents, or research and ED staff. The children and their parents will be informed that the study is to evaluate different forms of distraction but will not know the study hypothesis for iPads nor what each group is receiving. The data analyst will be blind to treatment assignment through the use of randomization codes that will not be disclosed until analysis is complete.

Study Intervention and Comparison: The intervention will be the use of an iPad that will include a selection of child-appropriate games. We will select popular, age-appropriate items to include on the iPad, chosen based on the most current online consumer ratings. Children and parents will be able to select their choice of distraction and can change their selection as desired during the course of the procedure. These choices will be recorded for study purposes. The control group will receive standard care, which generally includes the use of topical anesthetic cream. This comparison is based on the pragmatic preferences of physicians at the Stollery Children's Hospital as well as precedent in the literature. Overall, it is felt that any new intervention (e.g., iPad) should be compared to what is currently in practice (i.e., standard care), as no single distraction therapy is consistently and routinely employed in EDs at this time.

Study Outcomes: The primary outcomes are patient pain and distress. Self-reported pain will be measured using the Faces Pain Scale-Revised (FPS-R). This measurement will be made immediately following the initial attempt at IV placement. The FPS-R is the currently recommended pain scale for our participant group with strong evidence of validity and reliability for our age range. Distress will be measured using the Observed Scale of Behavioral Distress-Revised (OSBD-R); a tool designed to assess a child's behavioural response to painful medical procedures. The scale scores are reliable and valid for our target population. Two research students will be trained in the use of the tool and will independently observe a videotape of each child and record the frequency of operationally-defined distress-related behaviours during continuous 15-second intervals before, during, and after the procedure. This protocol for use of the OSBD-R is standard; it has been used in other trials evaluating distraction, including a trial by one of the PIs (LH) evaluating music. The secondary outcomes are (a) observed pain which will be measured by the research students using a standard 100 mm visual analogue scale; (b) parent and provider satisfaction (measured using Likert scales); (c) ease of performing the procedure assessed by the provider; time to complete the procedure; (d) success of the procedure; and (e) parent state anxiety measured with a validated instrument, the State Trait Anxiety Inventory (STAI-S, Form Y).

ELIGIBILITY:
Inclusion Criteria:

* attending pediatric emergency department
* require IV placement
* fully conscious and alert
* have sufficient knowledge of the English language to understand and complete the pain assessments

Exclusion Criteria:

* hearing or visual impairments
* neurocognitive delays
* sensory impairment to pain (e.g., spina bifida)
* at the discretion of the attending staff (e.g., child in critical condition)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
pain (self report) Faces Pain Scale-Revised (FPS-R) | at time of IV placement, Day 1
  Faces Pain Scale-Revised (FPS-R)
distress Observed Scale of Behavioral Distress-Revised (OSBD-R) | at time of IV placement, Day 1
  Observed Scale of Behavioral Distress-Revised (OSBD-R)

SECONDARY OUTCOMES:
pain (observed) visual analogue scale | at time of IV placement, Day 1
  measured by the research students using a standard 100 mm visual analogue scale
parent and provider satisfaction (Likert scale) | 2 minutes post IV placement, Day 1
  Likert scale
ease of procedure performance (assessed by provider) | at time of IV placement, Day 1
  assessed by provider
success of procedure (assessed by provider) | at time of IV placement, Day 1
  assessed by provider
parent anxiety (State Trait Anxiety Inventory (STAI-S, Form Y) | at time of IV placment, Day 1
  State Trait Anxiety Inventory (STAI-S, Form Y)

CONTACTS AND LOCATIONS:
Overall Officials: Samina Ali, MD, Principal Investigator — University of Alberta/Stollery Children's Hospital
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ali S, Ma K, Dow N, Vandermeer B, Scott S, Beran T, Issawi A, Curtis S, Jou H, Graham TAD, Sigismund L, Hartling L. A randomized trial of iPad distraction to reduce children's pain and distress during intravenous cannulation in the paediatric emergency department. Paediatr Child Health. 2020 Aug 20;26(5):287-293. doi: 10.1093/pch/pxaa089. eCollection 2021 Aug. PMID 34630780